CLINICAL TRIAL: NCT03407573
Title: The Impact of Restrictive Versus Liberal Transfusion Strategy on Cardiac Injury in Patients Undergoing Surgery for Fractured Neck Of Femur Study
Brief Title: Restrictive vs Liberal Transfusion Strategy on Cardiac Injury in Patients Undergoing Surgery for Fractured Neck Of Femur
Acronym: RESULT-NOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: WKRO-2016-0018
Record Dates: First submitted 2017-02-22; First posted 2018-01-23 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2018-03

CONDITIONS: Anemia; Cardiac Event; Kidney Injury; Fractured Hip
MeSH Terms: conditions — Anemia; Cardiovascular Diseases; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive (Active Comparator): Restrictive transfused when Hb at or below 70
  Interventions: Biological: Administration of Red Cell
- Liberal (Active Comparator): Will receive blood transfusion when Hb drops below or equal to 90
  Interventions: Biological: Administration of Red Cell

INTERVENTIONS:
Biological: Administration of Red Cell — Transfusion of red cells dependent on haemoglobin level. Either transfused at haemoglobin of 7 or 9.

SUMMARY:
The investigator wishes to see if it is possible to undertake a study comparing blood transfusion at two different levels of anaemia to see which is best for patients. All patients that present to hospital with a broken hip will be able to take part in the study. If they become anaemic during their treatment they will be allocated to either be transfused when their blood count is less that 9 or less than 7. In all patients, we will measure heart damage with a blood test that is very sensitive. The investigator will also collect data on the incidence of heart attacks and other complications.

DETAILED DESCRIPTION:
Many frail and elderly patients undergo surgery for hip fractures every year. Many of these patients have other health problems including heart disease and anaemia (low haemoglobin or "low blood count") either from chronic illness, from bleeding at the time of their injury or during subsequent surgery. The vast majority (more than 95%) of these patients will go on to have surgery. This surgery is often high risk. Patients with this type of injury may already be frail, may be in hospital for a long time and will need rehabilitation. Many of them will develop complications, including heart attacks and some will die.

Doctors looking after these patients commonly prescribe a blood transfusion around the time of surgery. These patient often have anaemia before surgery an lose more blood during their operations. A benefit of blood transfusion is that it may increase the amount of oxygen the blood can carry. One of the main reasons that doctors prescribe blood around the time of surgery is to prevent heart attacks, which can occur if the heart doesn't receive enough oxygen. Another possible benefit of blood transfusion is that it may help patients get out of bed more quickly after surgery. This is another important aspect of their recovery.

However, blood transfusions can have side effects such as causing heart failure or increasing infections after surgery. These can delay patient recovery too. Although some research has been done in this area, anaesthetists and surgeons are still unsure of when to prescribe blood transfusions to these patients. In particular, uncertainty about how low the blood count should be before a blood transfusion is ordered. Some doctors prescribe blood when the haemoglobin count is less than 9 and some at a lower level of 7. Current guidelines suggest that prescribing at a lower haemoglobin count is better, but there is research which suggests that this level is too low if the patient has a history of heart disease.

ELIGIBILITY:
Inclusion Criteria:Adults aged over 50 years Within 48 hours of admission to hospital with fractured Neck of Femur. Exclusion Criteria: Age <50

* Refusal of consent of patient (or consultee) Patient for palliative care.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Myocardial Injury | Upto 60 days
  Myocardial injury defined as a high sensitivity cardiac Troponin 1 (Troponin) concentration above the upper reference limit [URL] OF 16 ng L and 34 ng L in women and men respectively at any time during the study period.

SECONDARY OUTCOMES:
Myocardial Infarction | within 30 days of surgery
  Myocardial Infarction defined per the universal definition within 30 days of surgery or before hospital discharge, whichever occurs first.
Mortality | upto 60 days following surgery
  Mortality (30; 60 days from day of surgery).
Diagnosis of Major Adverse Cardiac Events | within 30 days or before hospital discharge
  New diagnosis of MACE within 30 days of surgery or before hospital discharge, whichever occurs first.
Acute Kidney Injury | within 30 days of surgery or before discharge from hospital whichever occurs first.
  New diagnosis of Acute Kidney Injury
Infections | within 30 days of surgery or before hospital discharge, whichever is first.
  New diagnosis of Infectious Complications
Delirium | within 30 days of surgery or before hospital discharge, whichever occurs first.
  New diagnosis of Delirium

OTHER OUTCOMES:
Troponin | within 7 days of surgery (ngL )
  Peak troponin concentration
Troponin -Time | within 7 days of surgery
  Area under a Troponin-Time curve
Red cells transfused | within7 days of surgery and within 30 days of surgery or before hospital discharge, whichever occurs first.
  Number of units red cells transfused
Volume in mls of Red Cells Transfused. | within 7 days of surgery and within 30 days of surgery or before hospital discharge, whichever occurs first.
  Volume of red blood cells transfused in mls
Haemoglobin postoperatively | days 1,3,5,7 after surgery
  Postoperative Hb on postoperative days
Nadir Hb | within 7 days of surgery and within 30 days of surgery or before hospital discharge, whichever occurs first.
  Nadir Hb
Hospital Admission | from admission to discharge date from hospital upto 60 days.
  Duration of hospital admission (days)
Readmission to hospital | upto 60 days of hospital discharge date
  Incidence of unplanned hospital readmission within 60 days
Destination | at Discharge from hospital with fractured hip upto 60 days of admission
  Discharge destination (home, other hospital, nursing home, other)
Health Related Quality of Life | at 60 days after surgery
  HRQoL at 60 days (EQ 5D)
Costs | 60 days post randomisation
  Secondary care costs during 60 days post-randomisation in Great British Pound

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mike Gillies, Principal Investigator — Associate Medical Director
Locations (1):
- Royal Hospital for Sick Children, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acheson AG, Brookes MJ, Spahn DR. Effects of allogeneic red blood cell transfusions on clinical outcomes in patients undergoing colorectal cancer surgery: a systematic review and meta-analysis. Ann Surg. 2012 Aug;256(2):235-44. doi: 10.1097/SLA.0b013e31825b35d5. PMID 22791100
- [Result] Fowler AJ, Ahmad T, Phull MK, Allard S, Gillies MA, Pearse RM. Meta-analysis of the association between preoperative anaemia and mortality after surgery. Br J Surg. 2015 Oct;102(11):1314-24. doi: 10.1002/bjs.9861. PMID 26349842
- [Result] Davenport DL, Bowe EA, Henderson WG, Khuri SF, Mentzer RM Jr. National Surgical Quality Improvement Program (NSQIP) risk factors can be used to validate American Society of Anesthesiologists Physical Status Classification (ASA PS) levels. Ann Surg. 2006 May;243(5):636-41; discussion 641-4. doi: 10.1097/01.sla.0000216508.95556.cc. PMID 16632998
- [Result] Holst LB, Petersen MW, Haase N, Perner A, Wetterslev J. Restrictive versus liberal transfusion strategy for red blood cell transfusion: systematic review of randomised trials with meta-analysis and trial sequential analysis. BMJ. 2015 Mar 24;350:h1354. doi: 10.1136/bmj.h1354. PMID 25805204
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Gillies MA, Ghaffar S, Moppett IK, Docherty AB, Clarke S, Rea N, Stephen J, Keerie C, Ray DC, White TO, MacLullich AMJ, Mills NM, Rowley MR, Murthy K, Pearse RM, Stanworth SJ, Walsh TS. A restrictive versus liberal transfusion strategy to prevent myocardial injury in patients undergoing surgery for fractured neck of femur: a feasibility randomised trial (RESULT-NOF). Br J Anaesth. 2021 Jan;126(1):77-86. doi: 10.1016/j.bja.2020.06.048. Epub 2020 Jul 21. PMID 32703548